CLINICAL TRIAL: NCT04742205
Title: Effectiveness of Intravenous Tranexamic Acid in Primary Cerebral Hemorrhage for Prevention of Hematoma Progression: Protocol for a Randomized, Double Blind Placebo-controlled Trial
Brief Title: ITCH Trial: Protocol for a Randomized, Double Blind Placebo-controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kathmandu Medical College and Teaching Hospital (Other)
Responsible Party: Principal Investigator, Bibesh Pokhrel, Lecturer, Kathmandu Medical College and Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KathmanduMCTH
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Hemorrhage
Keywords: double blind randomized trial; spontaneous intracerebral hemorrhage; tranexamic acid
MeSH Terms: conditions — Cerebral Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tranexamic acid (Active Comparator): Four 5ml solution of either tranexamic acid 500mg or sodium chloride 0.9% are distributed which cannot be differentiated from the appearance. Loading dose of trial (1g of tranexamic acid in 10ml) or placebo (10 ml of sodium chloride 0.9%) is mixed in 100ml sodium chloride 0.9% and given over 10 minutes. Maintenance dose of trial or placebo mixed in 500ml sodium chloride 0.9% is given over 8 hours
  Interventions: Drug: Tranexamic Acid 500 MG
- Sodium Chloride (Placebo Comparator): Four 5ml solution of either tranexamic acid 500mg or sodium chloride 0.9% are distributed which cannot be differentiated from the appearance. Loading dose of trial (1g of tranexamic acid in 10ml) or placebo (10 ml of sodium chloride 0.9%) is mixed in 100ml sodium chloride 0.9% and given over 10 minutes. Maintenance dose of trial or placebo mixed in 500ml sodium chloride 0.9% is given over 8 hours
  Interventions: Drug: Tranexamic Acid 500 MG

INTERVENTIONS:
Drug: Tranexamic Acid 500 MG — Loading dose of trial (1g of tranexamic acid in 10ml) is mixed in 100ml sodium chloride 0.9% and given over 10 minutes. Maintenance dose of trial mixed in 500ml sodium chloride 0.9% is given over 8 hours

SUMMARY:
Intracerebral hemorrhage is increasingly becoming a major burden in the society because of significant morbidity as well as mortality. Hematoma volume at the time of presentation as well as hematoma expansion and re-bleed or ongoing bleed further deteriorates the patient making a poor prognosis, however at present no therapy targets this pathological process. Though clinical studies do report benefit of using tranexamic acid in spontaneous intracerebral hemorrhage by reducing hematoma expansion rate as well as decreasing ongoing bleed, large randomized controlled trials have not shown any convincing advantage owing to various limitations in their design and methods. However, they uniformly did not find any significant side effect with the use of tranexamic acid.

The aim of this study is to test the hypothesis that intravenous tranexamic acid is superior to placebo by reducing hematoma expansion when given within 24 h of spontaneous intracerebral hemorrhage.

DETAILED DESCRIPTION:
Patients and Methods: Data are being collected as patient gets admitted with Intracerebral haemorrhage. 154 spontaneous intracerebral haemorrhage patients presenting within 24 hours of ictus or last known well will be taken in the study. Outcomes of these patients will be calculated to establish a relationship between hematoma expansion, underlying pathology and outcome of the patients.

Results: Primary outcome i.e. radiological improvement (CT scan): Difference between hematoma volume with perilesional edema from baseline and 48-hour post treatment scan, hematoma location, and new infarction.

Secondary outcomes: Neurological impairment (NIHSS), Disability (Barthel index), dependency (mRS) on day of discharge. mRS at day 30. Cognition (Telephone Interview Cognition Score-Modified), dependency (mRS) at days 90 and 180. Similarly, costs of treatment between two groups, length of stay in hospital and f/u data. Also, Safety endpoints recorded until day 180: Death (cause), venous thromboembolism confirmed by ultrasound, vascular occlusive events (stroke/transient ischemic attack/myocardial infarction/peripheral artery disease), seizures. Serious adverse events (AEs) in first seven days will be analyzed and calculated.

ELIGIBILITY:
Inclusion Criteria:

1. All patients presenting to the emergency department with symptom of hemorrhagic stroke within 24 hours from onset of symptom or last seen well.
2. Patient who had a follow up

Exclusion Criteria:

1. Glasgow coma scale <8 after resuscitation (as this can lead to biasness; requires surgery)
2. Contraindication to tranexamic acid,
3. Hemorrhagic stroke secondary to trauma,
4. Hemorrhage was caused by coagulopathy

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Radiological improvement (CT scan) | 48 hour
  Difference between hematoma volume from baseline and 48-hour post treatment scan

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale | day 10
  Neurological impairment (score:0-42; 0:favourable outcome)
Barthel index | days 10
  Disability (score:0-100; 100: independent)
modified rankin scale | days 10 and 30, 90, 180
  dependency (score:0-5; 0: no symptom)

OTHER OUTCOMES:
Death | day 180
  Number of death

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Regmi, MS, Study Chair — KMC AmbA
Locations (1):
- KMC Teaching Hospital, Kathmandu, Nepal, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Qureshi AI, Palesch YY, Barsan WG, Hanley DF, Hsu CY, Martin RL, Moy CS, Silbergleit R, Steiner T, Suarez JI, Toyoda K, Wang Y, Yamamoto H, Yoon BW; ATACH-2 Trial Investigators and the Neurological Emergency Treatment Trials Network. Intensive Blood-Pressure Lowering in Patients with Acute Cerebral Hemorrhage. N Engl J Med. 2016 Sep 15;375(11):1033-43. doi: 10.1056/NEJMoa1603460. Epub 2016 Jun 8. PMID 27276234
- [Background] van Asch CJ, Luitse MJ, Rinkel GJ, van der Tweel I, Algra A, Klijn CJ. Incidence, case fatality, and functional outcome of intracerebral haemorrhage over time, according to age, sex, and ethnic origin: a systematic review and meta-analysis. Lancet Neurol. 2010 Feb;9(2):167-76. doi: 10.1016/S1474-4422(09)70340-0. Epub 2010 Jan 5. PMID 20056489
- [Background] Dowlatshahi D, Demchuk AM, Flaherty ML, Ali M, Lyden PL, Smith EE; VISTA Collaboration. Defining hematoma expansion in intracerebral hemorrhage: relationship with patient outcomes. Neurology. 2011 Apr 5;76(14):1238-44. doi: 10.1212/WNL.0b013e3182143317. Epub 2011 Feb 23. PMID 21346218
- [Background] Brouwers HB, Greenberg SM. Hematoma expansion following acute intracerebral hemorrhage. Cerebrovasc Dis. 2013;35(3):195-201. doi: 10.1159/000346599. Epub 2013 Feb 28. PMID 23466430
- [Background] Steiner T, Bosel J. Options to restrict hematoma expansion after spontaneous intracerebral hemorrhage. Stroke. 2010 Feb;41(2):402-9. doi: 10.1161/STROKEAHA.109.552919. Epub 2009 Dec 31. PMID 20044536
- [Background] Flaherty ML, Haverbusch M, Sekar P, Kissela B, Kleindorfer D, Moomaw CJ, Sauerbeck L, Schneider A, Broderick JP, Woo D. Long-term mortality after intracerebral hemorrhage. Neurology. 2006 Apr 25;66(8):1182-6. doi: 10.1212/01.wnl.0000208400.08722.7c. PMID 16636234
- [Background] Zehtabchi S, Abdel Baki SG, Falzon L, Nishijima DK. Tranexamic acid for traumatic brain injury: a systematic review and meta-analysis. Am J Emerg Med. 2014 Dec;32(12):1503-9. doi: 10.1016/j.ajem.2014.09.023. Epub 2014 Sep 28. PMID 25447601
- [Background] Roos Y, Rinkel G, Vermeulen M, Algra A, van Gijn J. Antifibrinolytic therapy for aneurysmal subarachnoid hemorrhage: a major update of a cochrane review. Stroke. 2003 Sep;34(9):2308-9. doi: 10.1161/01.STR.0000089030.04120.0E. Epub 2003 Aug 21. No abstract available. PMID 12933970
- [Background] Germans MR, Post R, Coert BA, Rinkel GJ, Vandertop WP, Verbaan D. Ultra-early tranexamic acid after subarachnoid hemorrhage (ULTRA): study protocol for a randomized controlled trial. Trials. 2013 May 16;14:143. doi: 10.1186/1745-6215-14-143. PMID 23680226
- [Background] Mahmood A, Roberts I, Shakur H. A nested mechanistic sub-study into the effect of tranexamic acid versus placebo on intracranial haemorrhage and cerebral ischaemia in isolated traumatic brain injury: study protocol for a randomised controlled trial (CRASH-3 Trial Intracranial Bleeding Mechanistic Sub-Study [CRASH-3 IBMS]). Trials. 2017 Jul 17;18(1):330. doi: 10.1186/s13063-017-2073-6. PMID 28716153
- [Background] Anderson CS, Huang Y, Wang JG, Arima H, Neal B, Peng B, Heeley E, Skulina C, Parsons MW, Kim JS, Tao QL, Li YC, Jiang JD, Tai LW, Zhang JL, Xu E, Cheng Y, Heritier S, Morgenstern LB, Chalmers J; INTERACT Investigators. Intensive blood pressure reduction in acute cerebral haemorrhage trial (INTERACT): a randomised pilot trial. Lancet Neurol. 2008 May;7(5):391-9. doi: 10.1016/S1474-4422(08)70069-3. Epub 2008 Apr 7. PMID 18396107
- [Background] Arumugam A, A Rahman NA, Theophilus SC, Shariffudin A, Abdullah JM. Tranexamic Acid as Antifibrinolytic Agent in Non Traumatic Intracerebral Hemorrhages. Malays J Med Sci. 2015 Dec;22(Spec Issue):62-71. PMID 27006639
- [Background] Sprigg N, Flaherty K, Appleton JP, Al-Shahi Salman R, Bereczki D, Beridze M, Christensen H, Ciccone A, Collins R, Czlonkowska A, Dineen RA, Duley L, Egea-Guerrero JJ, England TJ, Krishnan K, Laska AC, Law ZK, Ozturk S, Pocock SJ, Roberts I, Robinson TG, Roffe C, Seiffge D, Scutt P, Thanabalan J, Werring D, Whynes D, Bath PM; TICH-2 Investigators. Tranexamic acid for hyperacute primary IntraCerebral Haemorrhage (TICH-2): an international randomised, placebo-controlled, phase 3 superiority trial. Lancet. 2018 May 26;391(10135):2107-2115. doi: 10.1016/S0140-6736(18)31033-X. Epub 2018 May 16. PMID 29778325
- [Background] Gayet-Ageron A, Prieto-Merino D, Ker K, Shakur H, Ageron FX, Roberts I; Antifibrinolytic Trials Collaboration. Effect of treatment delay on the effectiveness and safety of antifibrinolytics in acute severe haemorrhage: a meta-analysis of individual patient-level data from 40 138 bleeding patients. Lancet. 2018 Jan 13;391(10116):125-132. doi: 10.1016/S0140-6736(17)32455-8. Epub 2017 Nov 7. PMID 29126600
- [Background] O'Donnell MJ, Chin SL, Rangarajan S, Xavier D, Liu L, Zhang H, Rao-Melacini P, Zhang X, Pais P, Agapay S, Lopez-Jaramillo P, Damasceno A, Langhorne P, McQueen MJ, Rosengren A, Dehghan M, Hankey GJ, Dans AL, Elsayed A, Avezum A, Mondo C, Diener HC, Ryglewicz D, Czlonkowska A, Pogosova N, Weimar C, Iqbal R, Diaz R, Yusoff K, Yusufali A, Oguz A, Wang X, Penaherrera E, Lanas F, Ogah OS, Ogunniyi A, Iversen HK, Malaga G, Rumboldt Z, Oveisgharan S, Al Hussain F, Magazi D, Nilanont Y, Ferguson J, Pare G, Yusuf S; INTERSTROKE investigators. Global and regional effects of potentially modifiable risk factors associated with acute stroke in 32 countries (INTERSTROKE): a case-control study. Lancet. 2016 Aug 20;388(10046):761-75. doi: 10.1016/S0140-6736(16)30506-2. Epub 2016 Jul 16. PMID 27431356
- [Background] Antihypertensive Treatment of Acute Cerebral Hemorrhage (ATACH) investigators. Antihypertensive treatment of acute cerebral hemorrhage. Crit Care Med. 2010 Feb;38(2):637-48. doi: 10.1097/CCM.0b013e3181b9e1a5. PMID 19770736
- [Derived] Eilertsen H, Menon CS, Law ZK, Chen C, Bath PM, Steiner T, Desborough MJ, Sandset EC, Sprigg N, Al-Shahi Salman R. Haemostatic therapies for stroke due to acute, spontaneous intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD005951. doi: 10.1002/14651858.CD005951.pub5. PMID 37870112